CLINICAL TRIAL: NCT02706912
Title: Virtual Occupational Therapy Application
Acronym: VOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOTA1
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Hemiparesis; Activities of Daily Living; Virtual World; Occupational Therapy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VOTA Group (Experimental): All enrolled subjects are in this arm. After pre-assessment subjects have an 8-week waiting period, after which a mid-assessment takes place. Subject then participate in VOTA therapy for 8 weeks, followed by a post-assessment . The pre-/mid-assessment difference is used to control for spontaneous recovery. The mid-/post-assessment difference is used to ascertain efficacy.
  Interventions: Behavioral: VOTA Therapy

INTERVENTIONS:
Behavioral: VOTA Therapy — During sessions of approximately one hour in duration, participants practice performing virtual activities of daily living (ADLs) using the VOTA system. During this practice, the participant's real-world motion is replicated by an avatar's motion in the virtual world. To complete the activities, participant's must perform a wide range of functional arm movements while interacting with virtual objects. Individuals are asked to perform three such one-hour virtual ADL practice sessions per week over a participation period of approximately eight weeks.

SUMMARY:
Virtual Occupational Therapy Application (VOTA) combines low-cost human motion tracking, commercial game engine technology, and evidence-based Occupational Therapy (OT) practice in a computer-based virtual world in which stroke patients practice activities of daily living (ADLs). The protocol investigates the efficacy of VOTA therapy for Upper Extremity (UE) motor recovery and assesses system usability and user acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a hemiparetic stroke survivor;
* Time since last stroke at least 3 months;
* Participant has antigravity strength at the elbow to at least 45 degrees of active flexion in the stroke affected arm;
* Participant has antigravity shoulder strength to at least 30 degrees each in active flexion, abduction/adduction, and 15 degrees in active rotation from an upright seated position in the stroke affected arm;
* Participant has visual acuity with corrective lenses of 20/50 or better;

Exclusion Criteria:

* Existing participation in an upper extremity stroke rehabilitation program or planned participation during the study period;
* Inability to understand and follow verbal directions;
* Determination that participation would result in over exertion or significant discomfort or pain;
* Determination that participation would result in significant agitation or elevated stress;
* Withholding or withdrawal of consent by the participant;
* Visual field deficit in either eye that impairs the ability to view the computer monitor;
* Hemispatial neglect that impairs the ability process and perceive visual stimuli provided through the computer monitor;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity assessment | Pre-assessment and Post-assessment (8 weeks)
  Measure of upper extremity motor function

SECONDARY OUTCOMES:
Wolf Motor Function Test | Pre-assessment and Post-assessment (8 weeks)
  Measure of upper extremity motor function
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Pre-assessment and Post-assessment (8 weeks)
  Cognitive assessment
Trail Making Test | Pre-assessment and Post-assessment (8 weeks)
  Cognitive assessment

CONTACTS AND LOCATIONS:
Locations (1):
- UVA- HealthSouth Rehabilitation Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No